CLINICAL TRIAL: NCT06377657
Title: METRNL Response, Plasma Oxidative and Antioxidant Indices to HIIT and Aloe Vera Supplementation in Patients With Diabetes Type 2
Brief Title: Oxidative and Antioxidant Indices to HIIT and Aloe Vera Supplementation in Patients With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nis (Other)
Responsible Party: Principal Investigator, Anja Lazić, Junior Researcher, University of Nis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DONT4GET
Record Dates: First submitted 2024-03-23; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Type 2
Keywords: exercise, blood glucose oxidative stress, diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants were blinded for the supplementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-Intensity Interval Training (Experimental): Participants in HIIT group underwent 3 sessions per week for 12 weeks. The HIIT protocol (maximum 60 cycles per 20-minute session) includes 8-second fast pedaling (approximately 80% of maximum heart rate (HR max)) followed by slow pedaling (20-30 rpm) for 12 seconds. To facilitate acceleration and limit the stagnation of the bicycle wheel, the selected resistance was very low (almost zero).
  Interventions: Behavioral: Exercise
- Aloe Vera supplementation (Experimental): Participants in Aloe Vera group underwent supplementation with Aloe vera capsule containing 100 mg of Aloe vera gel powder in the morning immediately after waking up and one capsule after dinner.
  Interventions: Dietary Supplement: Aloe vera
- HIIT + Aloe Vera (Experimental): Participants in HIIT group underwent 3 sessions per week for 12 weeks. The HIIT protocol (maximum 60 cycles per 20-minute session) includes 8-second fast pedaling (approximately 80% of maximum heart rate (HR max)) followed by slow pedaling (20-30 rpm) for 12 seconds. To facilitate acceleration and limit the stagnation of the bicycle wheel, the selected resistance was very low (almost zero). Additionally, patients underwent supplementation with Aloe Vera capsules in the morning and after the dinner.
  Interventions: Behavioral: Exercise; Dietary Supplement: Aloe vera
- Control group (No Intervention): The control group continued their daily life activities for 12 weeks

INTERVENTIONS:
Behavioral: Exercise — The HIIT group underwent intervention with high intensity interval training. The second group was treated only with aloe vera supplementation for 12 weeks. A third group underwent a combination of HIIT and supplementation, while a fourth - CON group kept usual activities during the intervention duratino
  Arms: HIIT + Aloe Vera; High-Intensity Interval Training
Dietary Supplement: Aloe vera — Aloe Vera group was treated only with aloe vera supplementation for 12 weeks.
  Arms: Aloe Vera supplementation; HIIT + Aloe Vera

SUMMARY:
Diabetes is a prevalent metabolic disease that leads to increased blood sugar levels due to insulin shortage or resistance. Type 2 diabetes is often linked to obesity, which can increase insulin resistance. Meteorin-like protein (METRNL) is a new secreted protein that affects insulin sensitivity and has been found to be negatively related to serum glucose levels in people with diabetes.

Oxidative stress in diabetics can stimulate the production of inflammatory mediators, increasing the activity of the antioxidant system. Aloe vera, a widely used plant, has been used for treating diabetes, wound healing, tumors, and inflammatory bowel disease. It has anti-inflammatory, antioxidant, neuroprotective, antidepressant, and memory-enhancing effects.

Exercise can improve diabetic patients' conditions by increasing the expression of GLUT4 protein and skeletal muscle. High-intensity interval training has been shown to increase the expression of the METORIN gene in human subjects and decrease MDA in type 2 diabetic patients. However, no studies have examined the simultaneous effect of exercise and Aloe vera on diabetes indicators.

The present study aims to investigate the response of METRNL and some oxidative and antioxidant plasma indicators to high-intensity interval training and Aloe vera supplementation in type 2 diabetic men. The findings indicate that exercise and consumption of plants with anti-inflammatory and antioxidant properties can be effective in modulating the pathological effects of diabetes and increasing insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who have been diagnosed with T2DM at least 3 months prior to the start of the study according to standard criteria
* Inactive participants according to the International Physical Activity Questionnaire (IPAQ)
* Participants receiving stable medical therapy for T2DM, excluding those on exogenous insulin therapy
* Participants who were free from injuries or chronic health conditions that could limit their ability to safely participate in an intense exercise program were included in the study

Exclusion Criteria:

* Fasting glucose above 270 mg / dL
* Exogenous insulin
* History of diabetic complications (the final stage of proliferative diabetic retinopathy, or subsequent overt nephropathy, diabetic ketoacidosis, or severe diabetic neuropathy)
* Hereditary glucose and galactose malabsorption

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
METRNL - Meteorin Like, Glial Cell Differentiation Regulator | Baseline and 12 weeks
  Plasma METRNL content was measured using a special kit (Mybiosource company, USA) with a sensitivity of <0.64 ng / ml, range of 1.56-100 ng / ml by ELISA method

SECONDARY OUTCOMES:
Glutathione peroxidase (GPx) | Baseline and 12 weeks
  GPx was measured using a special kit (abcam company, USA) through ELISA method.
Serum superoxide dismutase (SOD) | Baseline and and 12 weeks
  SOD was measured using a special kit (Abcam company, USA) through ELISA method.
Total antioxidant blood capacity (TAD) | Baseline and 12 weeks
  TAD was measured using a special kit (Abcam company, USA) through ELISA method.
Plasma malondialdehyde (MDA) | Baseline and 12 weeks
  MDA was measured using a special kit (Abcam company, USA) through ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Lazić, Prof., Principal Investigator — Faculty of Sport and Physical Education, University of Niš
Locations (1):
- Department of Sport Physiology, Faculty of Sport and Physical education, Islamic Azad University of Ayatollah Amoli, Amol, Iran, Āmol, Iran